CLINICAL TRIAL: NCT06351865
Title: A Feasibility Study to Evaluate if Breast Cancer Patients, Consented Using Digital Consent, Reliably Provide Accurate Patient Reported Complication (PRC) Data Using Feedback Questionnaires
Brief Title: Feasibility Study to Evaluate the Use of Patient Reported Complications After Digital Consent
Acronym: PRC
Status: Recruiting | Type: Observational
Sponsor: Portsmouth Hospitals NHS Trust (Other Government)
Collaborators: University of East Anglia (Other)
Responsible Party: Sponsor
Other Study IDs: PHU/2023/21
Record Dates: First submitted 2024-04-02; First posted 2024-04-08 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer; Complication of Surgical Procedure
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patient report complication data to our best knowledge has not been studied yet in electronic consent. This study is a feasibility study to assess whether patients will reliably report their complications, the quality of this reporting and whether the information provided in the consent form matches up to their experience. This data will then be used to improve the consent process and evaluate whether the Patient Initiated Follow Up (PIFU) model is effective or if it leads to underreporting of problems.

DETAILED DESCRIPTION:
At the time of consent, patients are informed of possible post-operative complications. It is often not known whether these complications actually occur, whether there are others which go unreported and the extent, both quantitatively and qualitatively, of the complications. Patient reported complication data, to our best knowledge has not been previously studied.

This study is a feasibility study to assess whether patients will reliably report their complications, the quality of this reporting and whether the information provided in the consent form matches up to their experience. In this case, consent is to be sought digitally; the digital consent form includes a procedure specific list of recognised complications but these might not reflect actual patient experience.

If PRC data collection is feasible and reliable, this technique could be scaled to create a consent feedback loop, enabling operative outcome data to be collected from all patients, to be be used to improve the consent process for subsequent patients.

Awareness of post-operative patient complications is important and it is an NHS (National Health Service) requirement that complications are discussed within regular clinical governance (mortality/morbidity) audit departmental meetings. Currently this process relies on clinicians obtaining and reporting these complications. The move towards Patient Initiated Follow Up (PIFU) models may be leading to underreporting of problems. Potentially Patient Reported Complications would allow for a more comprehensive understanding of the benefits and consequences of the various surgical procedures. This in turn might help facilitate 'shared decision making' and allow treatment decisions to be tailored to the individual patients.

ELIGIBILITY:
Inclusion Criteria:

* Consent form 1- Adult patients who have the capacity to consent for themselves.
* Female adult aged 18years or above
* Diagnosed with early invasive breast cancer suitable for breast conserving surgery
* Undergoing Wide Local Excision of the breast and sentinel lymph node biopsy.
* Participant must be able to fill out an electronic questionnaire or take part in a phone questionnaire.
* Participant is willing and able to give informed consent for participation in the study.

Exclusion Criteria:

* Unable to consent for themselves or do not wish to participate.
* Patients who need an interpreter.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women over 18yrs old with early invasive breast cancer who are undergoing "wide local excision and sentinel lymph node biopsy" operation.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-03-07 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients who respond to the feedback questionnaire | 6 months
  Calculate the proportion of patients who respond to the feedback questionnaire
Final attrition rate | 6 months
  Calculate the final attrition rate. This is the proportion of patients who fail to respond to the email questionnaire and telephone call.

SECONDARY OUTCOMES:
Quoted risks in the consent to the incidence of complications | 6 months
  Compare the quoted risks in the consent to the incidence of complications reported by the patients.
Frequency of PRC and CRCs (Consent Form Reported Complications) | 6 months
  Review the monthly department CGM (Clinical Governance Meeting) data for the study period and correlate the frequency of PRC and CRCs.
Understanding of consent | 6 months
  Calculate the proportion of patients that feedback that they have understood the consent form.
Language used in patient reported complications | 6 months
  Examine the language used by patients in the free-text box for reporting complications and whether this matches to that use in their consent form.
Accuracy of potential complications | 6 months
  To examine the feedback from the patient questionnaire which asks, if they experienced a complication, was it mentioned as a possibility in their consent form.
Participant preparation for surgery | 6 months
  From the feedback from the patient questionnaire, do patients feel fully informed about the procedure they are undertaking and feel well prepared

CONTACTS AND LOCATIONS:
Overall Officials: Edward St John, Principal Investigator — Portsmouth Hospitals NHS Trust
Locations (1):
- Queen Alexandra Hospital, Portsmouth, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No